CLINICAL TRIAL: NCT06378762
Title: Interference of Endurance Training on Strength Development and Neuromuscular Adaptations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Miguel Gomes, Invited Assistant Professor, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6/2021
Record Dates: First submitted 2024-04-08; First posted 2024-04-22 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Exercise
Keywords: Neuromuscular adaptations; Concurrent training; Interference effect; Endurance; Strength
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Endurance (Experimental)
  Interventions: Behavioral: Endurance Exercise
- Strength (Experimental)
  Interventions: Behavioral: Strength Exercise
- Concurrent (Experimental)
  Interventions: Behavioral: Concurrent Exercise

INTERVENTIONS:
Behavioral: Endurance Exercise — 30 minutes of running at an intensity corresponding to the heavy-domain (between the first and second ventilatory thresholds)
  Arms: Endurance
Behavioral: Strength Exercise — Combination of strength and power exercises Weeks 1-5 focus on building maximal strength Weeks 6-11 focus on maintaining maximal strength and improve muscle power
  Arms: Strength
Behavioral: Concurrent Exercise — Combining both strength and endurance training programs, with strength preceding endurance, incorporating a 20-min rest period between each modality
  Arms: Concurrent

SUMMARY:
This study aims to find out if performing combined strength and endurance exercise in the same program (called concurrent training-CT) leads to similar long-term improvements in neuromuscular function as doing each type of exercise separately. The main questions it seeks to answer are:

Does performing CT result in similar improvements in strength and power as doing just strength training? Does performing CT result in similar improvements in cardiorespiratory fitness as doing just endurance training? Are neuromuscular adaptations similar between CT and just strength training? Researchers will compare the results between three groups: the CT group, the endurance training group (E), and the strength training group (S) to answer these questions.

DETAILED DESCRIPTION:
This study looks at how different types of exercise affect neuromuscular and cardiorespiratory improvements over time. It aims to see how combining strength and endurance training (concurrent training - CT) affects neuromuscular and cardiorespiratory adaptations compared to doing just strength or endurance training. Participants who regularly do both types of exercise will be split into three groups: Concurrent training (CT), endurance training (E), or strength training (S) and will be involved in 11 weeks of supervised training, three days a week:

Endurance training involves 30 minutes of continuous running, three days a week, at an intensity corresponding to the heavy domain (between the first and second ventilatory threshold) Strength training includes weightlifting three days a week, focusing on building both strength and power.

Concurrent training incorporates both strength and endurance exercises in the same session, three days a week, with strength training being executed prior to endurance training.

Researchers will collect data at three time-points during the 11 weeks: before starting the program (Baseline), at the end of week 5 (Week 5), and at the end of the program (Week 11). Measurements include lower-body strength and power, aerobic capacity, nerve evoked responses, and muscle structure if the quadriceps femoris.

Researchers will then compare the CT, E, and S groups at each measurement point to see which type of training elicited the best adaptations for the different neuromuscular and cardiorespiratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Active training status (strength and endurance (running) exercise at least 2 times per week over the last three months prior to inclusion in the study)

Exclusion Criteria:

* Active smoking status
* Orthopedic injuries
* On medication
* Known cardiovascular or respiratory disease

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Maximal Isometric Strength | Baseline, Week 5, Week 11
  Maximal voluntary isometric strength of the plantarflexors and leg press exercise in Newtons
Maximal Dynamic Strength | Baseline, Week 5, Week 11
  Maximal dynamic strength on the back squat exercise in kilograms lifted
Surface EMG | Baseline, Week 5, Week 11
  Using surface electromyography (EMG), the muscle activation of the plantarflexors muscles will me assessed, as well as the quadriceps femoris during the leg press and back squat exercise
H-reflex excitability | Baseline, Week 5, Week 11
  Using percutaneous electrostimulation of the tibial nerve, spinal reflex excitability will be explored by assessing H-reflex evoked responses
V-wave | Baseline, Week 5, Week 11
  Using percutaneous electrostimulation of the tibial nerve, neural drive to the active muscle will be assessed by measuring V-wave amplitudes
Lower Body Muscle Power | Baseline, Week 5, Week 11
  Lower body muscle power in watts will be assessed during countermovement jumps
Muscle fascicle length | Baseline, Week 5, Week 11
  Fascicle length of the vastus lateralis muscles in centimeters
Muscle fascicle pennation angle | Baseline, Week 5, Week 11
  Pennation angle of the vastus laterais fascicles, in degrees
Muscle thickenss | Baseline, Week 5, Week 11
  Muscle thickenss of the vastus lateralis, in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Motricidade Humana - Universidade de Lisboa, Lisbon, Cruz Quebrada - Dafundo, Portugal

IPD SHARING:
Plan to Share IPD: No